CLINICAL TRIAL: NCT00597870
Title: Physician-Sponsored IDE for the Talent Endoluminal Stent Graft System for the Treatment of Thoracic Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rodney A. White, M.D. (Other)
Responsible Party: Sponsor-Investigator, Rodney A. White, M.D., Chief, Vascular Surgery, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10837-01
Record Dates: First submitted 2007-12-28; First posted 2008-01-18 (Estimated); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-06

CONDITIONS: Thoracic Aortic Aneurysms; Thoracic Transections; Intramural Hematoma; Pseudoaneurysm; Thoracic Aortic Dissection
Keywords: TAA
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aneurysm, False; Dissection, Thoracic Aorta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment of Thoracic Lesions (Experimental): Endoluminal treatment of thoracic lesions
  Interventions: Device: Endoluminal treament of thoracic lesions

INTERVENTIONS:
Device: Endoluminal treament of thoracic lesions — Endoluminal treament of thoracic lesions with a thoracic stent-graft

SUMMARY:
The primary objective of this trial is to determine whether the Talent Thoracic Stent Graft, an investigational device, is a safe and effective method of treating thoracic aortic aneurysms (abnormal ballooning of the vessel wall) and other thoracic lesions (dissections, transections, pseudoaneurysms, penetrating ulcers, etc.). The endovascular method is a substitute for the major operation that is performed to treat the lesions.

DETAILED DESCRIPTION:
The endovascular method consists of the insertion of catheters (vinyl tubes) into both groin arteries. These catheters then allow positioning of artificial tubes or stent graft(s) into the diseased blood vessel without the need for major surgery which involves opening the chest. The blood vessel problem (thoracic aortic aneurysm/lesion) will be treated using an artificial bypass tube (stent graft) that will be placed inside the diseased artery. The stent graft(s) that will be used are made of polyester graft fabric sewn to a self-expanding nickel-titanium (Nitinol) wire frame and is manufactured by Medtronic AVE, Santa Rosa California.

Aneurysms/lesions can be located in any position along the length of the aorta. This study evaluates only aneurysms/lesions that occur in the descending part of the thoracic aorta as it traverses the chest and enters the abdominal cavity. The risk of thoracic aneurysms/lesions is that they rupture without warning. The risk of rupture increases as the aneurysm size increases. Following rupture, almost all patients expire within the first 24 hours. For this reason treatment of thoracic aneurysms/lesions is recommended by conventional surgical means if the patient is a candidate for an operation. The conventional operation involves occluding the aorta and replacing the aneurysm with a cloth tube that is sewn to replace the diseased part of the aorta. The major surgery and occlusion of the aorta that is part of the conventional surgery is directly related to several complications that have been reported in the literature. In addition, many patients are too ill for conventional surgery due to concomitant illnesses.

After the procedure, the patient will be followed at regular intervals (pre-discharge, 1 month, 6 months, 12 months and every year thereafter for life) as part of the evaluation of the experimental treatment. During this time, the patient will have several tests performed to evaluate the function of the repair. The tests will include clinical examination, x-rays of the chest and spiral CT scan. The experimental part is the placement of the TALENT Stent-Graft System using the catheter (endovascular) methods. The risk of the experimental catheter bypasses is that the procedure may not be successful. In most cases, this would require a standard operation to repair the problem. Sometimes there are other risks such as injury to the vessels. Small pieces of diseased arteries may be dislodged which may require removal. Bleeding may occur from introduction sites, and rarely, infection may develop. If a catheter bypass is unsuccessful, there can be added discomfort because the procedure may last longer.

The benefits of the procedure are that the patient might avoid some of of the pain and discomfort associated with standard operations. Major surgery is avoided and hospital stay may be much shorter. Patients may be able to return to usual daily activities sooner. In addition, patients who are too high risk for conventional surgical treatment can have their aneurysm treated using the endovascular graft if their anatomy is appropriate

ELIGIBILITY:
Inclusion Criteria:

Subjects who participate in this study as study patients must fulfill the following criteria:

* Subject is > 18 years of age.
* Subject is not pregnant or lactating. Females of child-bearing potential must practice a reliable method of contraception.
* Subject is diagnosed with one of the following conditions of the descending thoracic aorta. All conditions must be verified by diagnostic imaging [ultrasonography, computed tomography (CT), magnetic resonance imaging (MRI) or angiography].

  * A true (i.e., atherosclerotic) supraceliac aneurysm (fusiform or saccular type) with or without a co-existing aortic dissection or penetrating aortic ulcer
  * Aortic dissection of DeBakey Type I or II (Stanford A, proximal) in the absence of an aneurysm; OR
  * Penetrating aortic ulcer in the absence of an aneurysm; OR
  * Traumatic transection; OR
  * Pseudoaneurysm - traumatic or degenerative (i.e., one that does not involve all layers of the vessel and is not atherosclerotic in origin).
* Subject's anatomy is suitable for placement of the Medtronic/Talent Stent-Graft, with a distinct proximal aneurysm neck of 10 mm or more in length and a distal aneurysm neck of at least 10 mm.
* Subject has a TAA that is dilated to > 5 cm in diameter, > 1.5 times the diameter of the adjacent native/non-aneurysmal aorta, or is symptomatic.
* Subject has a proximal and distal aortic neck diameter > 18 mm and < 42 mm.
* Subject has an arterial access site, either peripherally or via infrarenal abdominal aorta that is adequate for introduction of the stent-graft delivery system.
* Subject is competent to give informed consent.
* Subject will be available for the periodic follow-up (surveillance) after the procedure.

Exclusion Criteria:

* Subjects who would participate as study subjects and who fulfill any of the following criteria may not participate in this study:
* Subject has TAA with less than 10 mm proximal fixation length.
* Subject has an aneurysm that would require exclusion by the stent-graft of the segment of the aorta that gives rise to dominant spinal cord/intercostal arteries.
* Subject has a lesion that prevents delivery or expansion of the device.
* Subject has systemic infection, or is suspected of having systemic infection.
* Subject has a known mycotic aneurysm.
* Subject is not available or is not willing to come back for periodic follow-up (surveillance) after the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2002-05; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney A. White, M.D., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- LAC Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited over several years from patients in the hospital and referrals from other hospitals, providers and clinics in the area.
Pre-assignment Details: Participants treated
Groups:
- Endoluminal Treatment of Thoracic Lesions: Successful endoluminal treatment of thoracic lesion with a thoracic stent graft
Period: Overall Study
Arm/Group | Endoluminal Treatment of Thoracic Lesions
Started | 304
Completed | 304
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Number of participants treated
Groups:
- Number of Patients: Endoluminal treatment of thoracic aneurysm, dissection, pseudoaneurysm, aortic ulcer, transection and other thoracic lesion.
Arm/Group | Number of Patients
Number analyzed (Participants) | 304
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 304
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 125
  Not Hispanic or Latino | 179
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 70
  White | 199
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 304

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Endoluminal Treatment of Thoracic Lesion
Description: Evaluate the number of patients who had successful treatment of their thoracic lesion using the Medtronic Talent Endoluminal Stent Graft..
Time Frame: Throughout study completion, an average of 1 year
Population: Only 294 participants out of the 304 initial participants were assessed for this Outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Whose Thoracic Lesions Were Successfully Excluded and Treated: Evaluate the number of patients whose thoracic stent-graft was successful in preventing blood to flow into the blood vessels during the initial surgery.
Arm/Group | Participants Whose Thoracic Lesions Were Successfully Excluded and Treated
Number analyzed (Participants) | 294
Participants | 294

2. Secondary Outcome: Number of Participants With Successful Device Delivery and Deployment
Description: Evaluate the number of patients where the thoracic device was successfully delivered and deployed within the patients' thoracic lesion.
Time Frame: Throughout study completion, an average of 1 year
Population: Only 294 participants out of the initial 304 participants were assessed for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants With Successful Endoluminal Device Delivery and Deployment: The Medtronic endoluminal stent graft was delivered and implanted effectively appropriately within the blood vessel.
Arm/Group | Number of Participants With Successful Endoluminal Device Delivery and Deployment
Number analyzed (Participants) | 294
Participants | 269

ADVERSE EVENTS:
Time Frame: From treatment through 5 years
Groups:
- Exclusion of Thoracic Lesions: Successful endoluluminal exclusion/treatment of thoracic lesions
Arm/Group | Exclusion of Thoracic Lesions
All-Cause Mortality (participants affected / at risk) | 86/304
Serious Adverse Events (participants affected / at risk) | 107/304
Other Adverse Events (participants affected / at risk) | 4/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exclusion of Thoracic Lesions (N=304)
Endoleak (Vascular disorders) | 107 (107) — Leaks on the proximal or dial end or through the stent graft (Type1, 2, 3 endoleaks)
Aortic Dissection (Vascular disorders) | 7 (7) — Dissection of thoracic lesion outside of the treated lesion
Acute renal failure (Renal and urinary disorders) | 9 (9)
MI (Cardiac disorders) | 14 (14)
Stroke (General disorders) | 14 (14)
Infection (Surgical and medical procedures) | 8 (8)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Transient paralysis (General disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exclusion of Thoracic Lesions (N=304)
Hematoma (Surgical and medical procedures) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2002-03-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT00597870/Prot_000.pdf